CLINICAL TRIAL: NCT05744557
Title: Vapocoolant Analgesia for Breast Lymphoscintigraphy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: <75% accrued participants
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Gilero, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0454; NCI-2023-01629 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-02-15; First posted 2023-02-27 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- num Vapocoolant (Experimental): vapocoolant anesthetic spray (a spray that cools and numbs the skin) to control pain during minor surgical procedures (such as lancing boils, incisions, injections and IV placements) and minor sport injuries
  Interventions: Other: num Vapocoolant

INTERVENTIONS:
Other: num Vapocoolant — Spray will be administered for 4 to 6 seconds from a distance of 3 to 6 inches to desired sites of skin

SUMMARY:
To learn if applying vapocoolant anesthetic spray ("Nüm") on the surface of the intended injection site will reduce the pain/anxiety associated with breast injections.

DETAILED DESCRIPTION:
Primary Objectives:

1. Establish feasibility of topical vapocoolant in the setting of breast lymphoscintigraphy.
2. Demonstrate safety of topical vapocoolant in the setting of breast lymphoscintigraphy.

Secondary Objectives:

1. To assess patient pain intensity associated with the performance of breast lymphoscintigraphy.
2. To evaluate the attitude from patients about supporting the continued offering of topical vapocoolant in the breast lymphoscintigraphy clinic.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient undergoing asubareolar breast lymphoscintigraphy injection will be eligible.
* Age ≥18 years old
* Ability to understand and the willingness to sign a written informed consent document.
* Childbearing potential, lactating, pregnant women will be included.

Exclusion Criteria:

* Patients who have allergy or had prior hypersensitivity to either of the vapocoolants including 1,1,1,3,3 Pentafluoropropane and 1,1,1,2-Tetrafluoroethane.
* Patients with uncontrolled intercurrent illness (insulin dependent and non-insulin dependent diabetes)
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjit Tewari, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/57/NCT05744557/ICF_000.pdf